CLINICAL TRIAL: NCT07198750
Title: Effect of High-Intensity Pulsed Electromagnetic Field Therapy as a Bimodal Intervention for Analgesia and Strengthening in Older Adults With Knee Osteoarthritis: A Randomized Double-Blind Controlled Clinical Trial
Brief Title: "Bimodal vs Unimodal High-Intensity Pulsed Electromagnetic Field Therapy in Older Adults With Knee Osteoarthritis"
Acronym: HIPEMF-OAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Ana Lilia Villagrana Rodríguez, Physician Specialist, Department of Physical and Rehabilitation Medicine, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI-151-25
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis; Osteoarthritis; Osteo Arthritis of the Knee; Gonarthrosis
Keywords: High-Intensity Pulsed Electromagnetic Fields; HI-PEMF; Super Inductive System; Knee Osteoarthritis; Gonarthrosis; Geriatric Rehabilitation; Chronic Pain; Functional Mobility
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Two-arm parallel design: Group A receives HI-PEMF applied to the knee only (unimodal), while Group B receives HI-PEMF applied to both the knee and quadriceps (bimodal). Both groups also perform the same home-based exercise program.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were informed that the intervention would be applied to the lower limb without specifying the anatomical region. The HI-PEMF equipment produces no perceptible sensations, aiding participant blinding. Outcome assessors were independent and unaware of group assignment. Care providers administering the intervention were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Unimodal HI-PEMF (Experimental): Participants in Group A will receive high-intensity pulsed electromagnetic field therapy (HI-PEMF) applied exclusively to the symptomatic knee (femorotibial joint) for 10 minutes per session, twice a week over 5 weeks, completing a total of 9 sessions. The intervention will use the "Chronic Pain" protocol of the BTL-6000 Super Inductive System. A standardized home-based exercise program will be provided to all participants.
  Interventions: Device: HI-PEMF - Knee (Chronic Pain Protocol); Behavioral: Home-Based Exercise Program
- Group B - Bimodal HI-PEMF (Experimental): Participants in Group B will receive high-intensity pulsed electromagnetic field therapy (HI-PEMF) applied to both the symptomatic knee (femorotibial joint) and the quadriceps muscle (rectus femoris), with 10 minutes per site, twice a week over 5 weeks, completing a total of 9 sessions. The knee application will follow the "Chronic Pain" protocol, and the quadriceps application will follow the "Muscle Strengthening" protocol, both using the BTL-6000 Super Inductive System. A standardized home-based exercise program will be provided to all participants.
  Interventions: Device: HI-PEMF - Quadriceps (Muscle Strengthening Protocol); Behavioral: Home-Based Exercise Program

INTERVENTIONS:
Device: HI-PEMF - Knee (Chronic Pain Protocol) — High-intensity pulsed electromagnetic field (HI-PEMF) therapy applied to the symptomatic knee using the "Chronic Pain" protocol of the BTL-6000 Super Inductive System, 10-minute duration per session, applied twice per week over 5 weeks (total of 9 sessions). The applicator is positioned 2-3 cm above the patella, without skin contact, with the patient seated or in supine position.
  Arms: Group A - Unimodal HI-PEMF
Device: HI-PEMF - Quadriceps (Muscle Strengthening Protocol) — HI-PEMF therapy will be applied to both the symptomatic knee and the quadriceps muscle (rectus femoris). The knee application will follow the same procedure as in Group A, using the "Chronic Pain" protocol of the BTL-6000 Super Inductive System. In addition, the quadriceps will be treated using the "Muscle Strengthening" protocol. Each site will receive 10 minutes of therapy per session, twice per week over 5 weeks (total of 9 sessions). The applicator for the quadriceps will be positioned perpendicular to the muscle belly, without skin contact, with the patient lying supine and a cushion under the knee for slight flexion.
  Arms: Group B - Bimodal HI-PEMF
Behavioral: Home-Based Exercise Program — Standardized home-based exercise program prescribed to both groups. It includes five exercises: isometric quadriceps contractions, straight leg raises, seated knee extensions, sit-to-stand from chair, and stationary marching. Participants are instructed to perform the exercises three times per week during the 5-week intervention. Printed instructions and a video guide are provided. Adherence is reinforced via weekly follow-up.

SUMMARY:
This randomized, double-blind clinical trial aims to evaluate the effect of high-intensity pulsed electromagnetic field therapy (HI-PEMF) applied either exclusively on the knee joint or bimodally on the knee and quadriceps, in older adults with knee osteoarthritis. Both groups will also receive a structured home-based exercise program. The primary outcome is pain reduction, and secondary outcomes include functional performance.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a highly prevalent and disabling condition in older adults. It often coexists with quadriceps muscle weakness, sarcopenia, and frailty, all of which contribute to pain, functional decline, and loss of independence. Pulsed electromagnetic field therapy (PEMF) has emerged as a non-invasive alternative for pain relief in OA, with growing interest in its application at both articular and muscular levels.

High-intensity pulsed electromagnetic field (HI-PEMF) therapy-also known as the super inductive system-generates magnetic fields up to 2.5 Tesla, capable of stimulating both joint structures and skeletal muscle via deep tissue electric induction. HI-PEMF has shown promising results for pain reduction, anti-inflammatory modulation, and muscle bioactivation, particularly when applied over the quadriceps.

This randomized, double-blind, parallel-assignment clinical trial aims to compare the effects of two HI-PEMF treatment modalities in older adults with moderate to severe knee OA (Kellgren-Lawrence grade II-IV):

* Group A: HI-PEMF applied exclusively over the symptomatic knee.
* Group 2: HI-PEMF applied both over the knee and the quadriceps (bimodal). Both groups will also perform a standardized home-based strengthening and mobility exercise program.

A total of 64 participants (32 per group) will receive 9 sessions of HI-PEMF (2 per week for 5 weeks), using the BTL-6000 Super Inductive System. Outcomes will be assessed at baseline and post-intervention. The primary outcome is change in pain intensity using the Numeric Analog Scale (NAS). Secondary outcomes include functional tests (Timed Up and Go and 5-times Sit-to-Stand), and paracetamol use. Exploratory subgroup analyses will assess associations with frailty status (FRAIL), probable sarcopenia (SARC-F), and radiological OA grade.

This study seeks to generate evidence on the potential synergistic benefits of combining articular and muscular HI-PEMF therapy in geriatric rehabilitation. It is designed for implementation in a public hospital setting in Mexico, with minimal risk and high feasibility. All procedures follow ethical guidelines and have received institutional review board approval.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60
* Clinical and radiological diagnosis of knee OA grade I-IV
* Pain ≥ 3 on Numeric Analog Scale for >6 months
* Can walk (with/without aid)
* Cognitive ability to follow instructions
* Signed informed consent
* Availability for 9 treatment sessions and home exercise Exclusion Criteria
* Prior total knee arthroplasty (unilateral or bilateral)
* Neurological disorders affecting motor function or cognition (e.g., Parkinson's disease, stroke, moderate to severe dementia)
* Active inflammatory rheumatic diseases (e.g., rheumatoid arthritis, lupus)
* Presence of pacemakers, implantable defibrillators, or metallic implants near the treatment area
* Current use of other physical therapy modalities for pain (e.g., electrotherapy, ultrasound, TENS) outside the study protocol
* Participation in another clinical trial within the past 3 months
* Current use of NSAIDs or systemic/local corticosteroids (including intra-articular injections)
* Open wounds or active infections at the treatment site
* Decompensated cardiac conditions or medical contraindication to exercise
* Vestibular disorders that affect balance and interfere with functional assessments
* Uncorrected visual impairment interfering with gait or balance (visual acuity worse than 20/60 in the better eye, assessed by Snellen chart)

Withdrawal Criteria:

* Participants who complete fewer than 7 out of the 9 planned intervention sessions (i.e., less than 80% adherence)
* Occurrence of serious adverse events related to the intervention that contraindicate continuation
* Repeated non-compliance with the home exercise program, documented in at least two consecutive weekly follow-up reports
* Voluntary withdrawal of consent at any time during the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity measured by the Numeric Analog Scale (NAS) | Baseline, end of intervention (week 5), and 2-month follow-up
  Pain intensity will be assessed using the 11-point Numeric Analog Scale (0 = no pain, 10 = worst possible pain), reported by the patient at rest and related to the most symptomatic knee. The primary endpoint is the change in NAS score from baseline to end of the 5-week intervention and at 2-month follow-up (approximately week 13). This will allow evaluation of both immediate and sustained effects of the intervention.

SECONDARY OUTCOMES:
Change in functional mobility measured by the Timed Up and Go (TUG) test | Baseline, end of intervention (week 5), and 2-month follow-up
  Functional mobility will be assessed using the Timed Up and Go (TUG) test. Participants are instructed to stand up from a chair, walk 3 meters, turn around, return, and sit down. The total time (in seconds) will be recorded using a stopwatch. The outcome measure is the change in time from baseline to the end of the 5-week intervention and at 2-month follow-up. This assesses both short-term and sustained improvements in functional mobility.
Change in lower-limb functional strength measured by the 5-times Sit-to-Stand (5STS) test | Baseline, end of intervention (week 5), and 2-month follow-up
  Lower-limb functional strength will be assessed using the 5-times Sit-to-Stand (5STS) test. Participants will be instructed to rise from a standard chair and sit back down five times as quickly as possible without using their arms. The total time (in seconds) to complete the task will be recorded using a stopwatch. The outcome measure is the change in time from baseline to the end of the 5-week intervention and at 2-month follow-up. This evaluates improvements in functional lower-limb strength and endurance over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared because the study is conducted within a public hospital setting without external funding, and there is no current plan or infrastructure to support secondary data sharing. Data will be used exclusively for the primary objectives outlined in the approved protocol.

REFERENCES:
- [Background] Iannitti T, Fistetto G, Esposito A, Rottigni V, Palmieri B. Pulsed electromagnetic field therapy for management of osteoarthritis-related pain, stiffness and physical function: clinical experience in the elderly. Clin Interv Aging. 2013;8:1289-93. doi: 10.2147/CIA.S35926. Epub 2013 Sep 26. PMID 24106421
- [Background] Ong MT, Man GC, Lau LC, He X, Qiu J, Wang Q, Chow MC, Choi BC, Yu M, Yung PS. Effect of pulsed electromagnetic field as an intervention for patients with quadriceps weakness after anterior cruciate ligament reconstruction: a double-blinded, randomized-controlled trial. Trials. 2022 Sep 12;23(1):771. doi: 10.1186/s13063-022-06674-2. PMID 36096886
- [Background] Bagnato GL, Miceli G, Marino N, Sciortino D, Bagnato GF. Pulsed electromagnetic fields in knee osteoarthritis: a double blind, placebo-controlled, randomized clinical trial. Rheumatology (Oxford). 2016 Apr;55(4):755-62. doi: 10.1093/rheumatology/kev426. Epub 2015 Dec 24. PMID 26705327